CLINICAL TRIAL: NCT01567111
Title: Functional Imaging With 11C-Metomidate Positron Emission Tomography Versus Adrenal Vein Sampling in Differential Diagnosis of Unilateral and Bilateral Aldosterone Secretion in Primary Aldosteronism
Brief Title: 11C-Metomidate PET Versus Adrenal Vein Sampling in Primary Aldosteronism
Acronym: MIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Turku University Hospital (Other Government); Tampere University (Other)
Responsible Party: Principal Investigator, Niina Matikainen, M.D., Ph.D., Specialist in endocrinology, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: T79/2011
Record Dates: First submitted 2012-03-26; First posted 2012-03-30 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Primary Hyperaldosteronism
Keywords: Primary aldosteronism; Aldosterone producing adenoma; Bilateral adrenal hyperplasia; Metomidate-Positron emission tomography
MeSH Terms: conditions — Hyperaldosteronism; Adrenocortical Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects with PA (Experimental): All study subjects have biochemically confirmed PA and undergo adrenal CT, AVS and MTO-PET to diagnose lateralization of aldosterone production.
  Interventions: Procedure: 11C-Metomidate Positron Emission Tomography

INTERVENTIONS:
Procedure: 11C-Metomidate Positron Emission Tomography — Dose of intravenous 11C-Metomidate injection is 440MBq and emission scanning of upper abdomen. PET/CT imaging will be done using the Discovery PET/CT VCT or 690 scanner (General Electric Medical Systems, Milwaukee, WI, USA)

SUMMARY:
Rationale: Primary hyperaldosteronism (PA) is the most frequent and possibly curable form of secondary hypertension. The diagnosis and targeted treatment of PA is essential because of high vascular morbidity associated with PA as compared to essential hypertension with comparable blood pressure levels. PA is usually caused by either a unilateral aldosterone-producing adenoma (APA) or by bilateral adrenal hyperplasia (BAH). Distinction between APA and BAH is critical since the former may be cured by adrenalectomy, and the latter needs life-long medical therapy with mineralocorticoid receptor antagonists (MRA). Studies demonstrate that adrenalectomy benefits also BAH patients with dominant nodule(s) producing the most of aldosterone excess. The distinction between unilateral and bilateral PA can be made by adrenal vein sampling (AVS), as recommended by The Endocrine Society 2008 guideline. Currently, in Finland the diagnosis is based on computed tomography (CT) scanning which does not distinguish between aldosterone-producing and common non-functioning adrenal nodules and has limited accuracy detecting small adrenal masses. Since AVS is invasive, dependent on skilled radiologist and costly, there is a need for an accurate, non-invasive functional imaging such as 11C-metomidate positron emission tomography (MTO-PET).

Objective: To assess diagnostic ability of MTO-PET as compared to AVS in PA. Secondary objectives: To compare if standardized uptake values (SUVs)in MTO-PET imaging are similar in histologically diagnosed nodular hyperplasia versus adenoma. To assess the diagnostic accuracy of adrenal CT as compared to MTO-PET and AVS. To assess the complete and partial remission rates (blood pressure response expressed in Daily Defined Dosages, medical therapy, use of potassium supplements) after allocating subjects to MRA-therapy or adrenalectomy at 1 and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Biochemically proven PA
* Good general health enabling possible adrenalectomy
* BMI less than 35

Exclusion Criteria:

* Any contraindication for AVS, MTO-PET or CT
* Subjects not willing to consider adrenal surgery
* Pregnancy
* Familial PA
* Suspicion of other tumor than adenoma or hyperplasia in adrenal CT scan

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-08 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Standard uptake value (SUV) in 11C metomidate Positron emission tomography (MTO-PET) | Up to 12 weeks
  Mean and maximun SUV-values detect lateralization / no lateralization in aldosterone production in MTO-PET as compared to AVS.

SECONDARY OUTCOMES:
Standard uptake value (SUV) in 11C metomidate Positron emission tomography (MTO-PET) | Up to 12 weeks
  Mean and maximun SUV-values detect lateralization / no lateralization in aldosterone production in MTO-PET as compared to adrenal CT.
Standard uptake value (SUV) in 11C metomidate Positron emission tomography (MTO-PET) | Up to 12 weeks
  Diffences between mean and maximum SUVs in MTO-PET between APA and BAH.
Blood pressure response | 1 and 5 years
  Daily Defined Dosages of hypertension medical therapy in subjects subjected to MRA or adrenalectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Niina Matikainen, M.D., Ph.D., Principal Investigator — Helsinki University Central Hospital
Locations (3):
- Finland (3):
  - Helsinki University Central Hospital, Helsinki
  - Tampere University, Tampere
  - University of Turku, Turku